CLINICAL TRIAL: NCT01097551
Title: Assessment of Endothelial Dysfunction in Retinal and Peripheral Retinal Vessels in Diabetes
Brief Title: Endothelial Dysfunction and Diabetes
Acronym: DENDI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P080608; 2009-A0109552 (Other: Eudra CT)
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Diabetic retinopathy; Pathogenesis; Dynamic Vessel Analyser; Endothelial dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy | interventions — Nitroglycerin; Phenylephrine; Iontophoresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with type 1 diabetes: Diabetes duration >= 5 years, age >= 18 and <= 60 years old, patients with no visible diabetic retinopathy, and no arterial hypertension
  Interventions: Drug: Trinitrin; Drug: Neosynephrine 10% collyrium; Drug: Iontophoresis with acetylcholine delivery; Device: Dynamic Vessel Analyzer
- Healthy subjects: Sex and age-matched control healthy subjects
  Interventions: Drug: Trinitrin; Drug: Neosynephrine 10% collyrium; Drug: Iontophoresis with acetylcholine delivery; Device: Dynamic Vessel Analyzer

INTERVENTIONS:
Drug: Trinitrin — Trinitrin: 2 sublingual pulverisations of 0.3 mg/dose
Drug: Neosynephrine 10% collyrium — Neosynephrine 10% collyrium: 2 drops
Drug: Iontophoresis with acetylcholine delivery — Iontophoresis with acetylcholine delivery
Device: Dynamic Vessel Analyzer — Dynamic Vessel Analyzer

SUMMARY:
The aim of the study is to progress in the understanding of the early retinal vascular and neural abnormalities in patients with diabetes, using a new device, the Dynamic Vessel Analyzer. The Dynamic Vessel Analyzer allows to measure the diameter of the retinal vessels and to assess how it varies in presence of various stimuli. Then, we will be able to assess if a vascular and/or a neural dysfunction is present early in patient with diabetes.

DETAILED DESCRIPTION:
Twenty patients with type 1 diabetes without diabetic retinopathy and without arterial hypertension will be compared with 20 sex and aged-matched healthy control subjects. To assess the presence of retinal endothelial dysfunction, the variations of the diameters of the retinal vessels will be assessed using the Dynamic Vessel Analyzer, before and after flicker light stimulation, sublingual nitroglycerin, neosynephrine eyedrops, and isometric contraction. To assess the presence of peripheral endothelial dysfunction, the microcirculation of the forearm skin will be studied using iontophoresis with acetylcholine delivery, and heat delivery, both coupled with blood flow measurement using laser Doppler. An intravital capillaroscopy of the phalanx skin will be performed. The serum levels of CRP, ICAM-1, VCAM-1, VEGF, angiopoietin 2 and endostatin will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* For diabetic patients :

  * age between 20 and 60
  * type 1 diabetes mellitus
  * diabetes duration of more than 5 years
  * no diabetic retinopathy on fundus examination or fundus photographs
  * no systemic hypertension (defined as systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
* For control subjects :

  * sex and age matching with the diabetic patients
  * no diabetes, no familial or personal history of elevated blood sugar
  * Non-diabetic subjects, criteria defined by a fasting glucose <1.10 g / l and an HbA1c <6.5% (according to Lariboisière biochemistry laboratory HbA1c)
  * no systemic hypertension (defined as systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
  * Subject with a normal ophthalmologic examination
* For both diabetic patients and control subjects :

  * Subject that has signed informed consent
  * Subject affiliated to a social security
  * Subject available for a period of 4 months

Exclusion Criteria:

* For both diabetic patients and control subjects :

  * presence of cataract or history of cataract surgery
  * intraocular pressure of more than 21 mmHg
  * treatment with vasoactive drugs
  * tobacco consumption of more than 20 cigarettes a day
  * Contraindications to trinitrin administration: hypersensitivity to trinitrin, treatment by sildenafil, heart disease, severe arterial hypotension, bradycardia, intracranial hypertension
  * Clinical Raynaud syndrome
  * Pregnant or breast-feeding subject
  * Subject whose age is <18 and> 60 years on the day of inclusion
  * Subject with cardiac disease, severe hypotension (BP <80/50 mmHg), a resting heart rate below 50 beats / minute
  * Subject intracranial hypertension
  * Subject with a current consumption of drugs or drugs that may impact vasomotion (antiglaucoma eye drops, vasodilators, antihypertensive drugs). Vasoactive drug use will be prohibited within 24 hours preceding the study.
  * Subject has not signed an informed consent
  * Subject not affiliated to a social security
  * Subject not available for a period of 4 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with type 1 diabetes: Diabetes duration >= 5 years, age >= 18 and <= 60 years old, patients with no visible diabetic retinopathy, and no arterial hypertension
  Healthy subjects: Sex and age-matched control healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the presence of a retinal endothelial dysfunction in patients with type 1 diabetes mellitus with Dynamic vessel analyser(assessment study visit) | up to 4 months

SECONDARY OUTCOMES:
Presence of a peripheral endothelial dysfunction | up to 4 months
Correlation between retinal and peripheral endothelial dysfunction (assessment study visit) | up to 4 months
Serum concentration of: CRP, ICAM-1, VCAM-1, VEGF, angiopoietin 2 and endostatin. | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Amélie LECLEIRE-COLLET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pascale MASSIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE Service d'Ophtalmologie, Paris, France